CLINICAL TRIAL: NCT03274141
Title: The Abatacept Best Care (ABC) Trial
Brief Title: Comparing the Effectiveness of a Treat-to-target (T2T) Disease Management Strategy vs. Routine Care (RC) in Adult Patients With Moderate to Severe Rheumatoid Arthritis (RA) Treated With Subcutaneous Abatacept (Orencia - SC)
Acronym: ABC
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-331
Record Dates: First submitted 2017-09-05; First posted 2017-09-06 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- T2T Patients: RA patients managed with a treat-to-target (T2T) strategy
  Interventions: Other: Non-Interventional
- RC Patients: RA patients managed with routine care(RC)
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
This is a 12 month prospective, multicenter, post-marketing, observational study to compare the effectiveness of a treat-to-target (T2T) disease management strategy vs. routine care (RC) in adult patients with moderate to severe rheumatoid arthritis (RA) treated with subcutaneous abatacept (Orencia - SC). Patients completing the study will be offered to participate in a 12-month extension of their follow-up provided that this is in agreement with the judgment of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Active moderate to severe RA, defined as CDAI > 10.
* The treating physician has made the decision to initiate treatment with SC abatacept in accordance with the Canadian product monograph.
* Patient has provided a written informed consent and is able to complete the survey requirements.
* Patient fulfills the reimbursement criteria for treatment with SC abatacept under provincial or private health insurance reimbursement coverage.

Exclusion Criteria:

* Has received abatacept (SC or IV) prior to the enrolment visit.
* Has failed more than one prior biologic DMARD therapy
* Has a history of autoimmune disease or of any joint inflammatory disease other than RA with the exception of concomitant secondary Sjogren's syndrome.
* Is participating in an ongoing clinical trial and/or has received treatment with an investigational agent within 4 weeks before starting treatment with SC abatacept.
* Is participating in another industry-sponsored observational study.
* Patients participating to non-industry related registries or other data collection studies can be included
* Presence of any condition that, in the opinion of the treating physician, prohibits the patient from participating in the study or obscures the assessment of RA treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with active RA defined as a CDAI > 10 for whom the treating physician has made the decision to initiate treatment with SC abatacept according to the approved Canadian product monograph and regional reimbursement criteria will be potentially eligible for inclusion in the study. The decision to treat the patient with SC abatacept must have been reached prior to and independently of considering the patient for study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Number of T2T patients achieving sustained CDAI LDA | Approximately 1 year
  Low Disease Activity (LDA) as determined by the Clinical Disease Activity Index (CDAI) is defined as a CDAI score of less than or equal to 10.
Number of RC patients achieving sustained CDAI LDA | Approximately 1 year
  Low Disease Activity (LDA) as determined by the Clinical Disease Activity Index (CDAI) is defined as a CDAI score of less than or equal to 10.

SECONDARY OUTCOMES:
Number of patients achieving SDAI remission | Up to 24 months
  Simplified Disease Activity Index (SDAI) remission is achieved when SDAI score is less than or equal to 3.3
Mean time for patients to achieve SDAI remission | Up to 24 months
  Length of time from treatment initiation SDAI remission
Number of patients achieving CDAI remission | Up to 24 months
  Clinical Disease Activity Index (CDAI) remission is achieved when CDAI score is less than or equal to 2.8
Mean time for patients to achieve CDAI remission | Up to 24 months
  Length of time from treatment initiation CDAI remission
Number of patients achieving DAS28-CRP LDA | Up to 24 months
  Disease Activity Score (DAS) Low Disease Activity (LDA) is achieved when DAS28-CRP score is less than 3.2
Mean time for patients to achieve DAS28-CRP LDA | Up to 24 months
  Length of time from treatment initiation to a DAS28-CRP score of less than 3.2
Number of patients achieving DAS28-CRP remission | Up to 24 months
  Disease Activity Score (DAS) remission is achieved when DAS28-CRP score is less than 2.6
Mean time for patients to achieve DAS28-CRP remission | Up to 24 months
  Length of time from treatment initiation to a DAS28-CRP score of less than 2.6
Number of patients achieving Boolean remission | Up to 24 months
  Boolean remission is defined as TJC28 ≤1 and SJC28 ≤1 and CRP ≤1 mg/dl and PtGA ≤1 (on a 0-10 scale)
Mean time for patients to achieve Boolean remission | Up to 24 months
  Length of time from treatment initiation to Boolean remission.
Number of patients achieving RAPID3 LDA | Up to 24 months
  Routine Assessment of Patient Index Data 3 (RAPID3) Low Disease Activity (LDA) is achieved when RAPID3 score is less than or equal to 6.
Mean time for patients to achieve RAPID3 LDA | Up to 24 months
  Length of time from treatment initiation to a RAPID3 score of less than or equal to 6
Number of patients achieving RAPID3 remission | Up to 24 months
  Routine Assessment of Patient Index Data 3 (RAPID3) remission is achieved when RAPID3 score is less than or equal to 3.
Mean time for patients to achieve RAPID3 remission | Up to 24 months
  Length of time from treatment initiation to a RAPID3 score of less than or equal to 3
Number of patients achieving MCID in HAQ-DI | Up to 24 months
  minimal clinically important difference (MCID; Δ ≥ 0.22, ≥0.25, and ≥0.5) in Health Assessment Questionnaire Disability Index (HAQ-DI)
Mean time for patients to achieve MCID in HAQ-DI | Up to 24 months
  Length of time from treatment initiation to a Δ ≥ 0.22, ≥0.25, and ≥0.5 in HAQ-DI
Number of patients achieving clinically meaningful improvement | Up to 24 months
  Number of patients achieving clinically meaningful improvement as measured by a decrease in CDAI of ≥ 20 or DAS28-CRP ≥ 1.2
Mean time for patients to achieve clinically meaningful improvement | Up to 24 months
  Length of time from treatment initiation to a decrease in CDAI of ≥ 20 or DAS28-CRP ≥ 1.2
Number of patients achieving patient expectations for treatment of their RA | Up to 24 months
  Assessed using simple Visual Analogue Scales (VAS)
Change from baseline in DAS28-CRP score | Baseline up to 24 months
  Measured by investigator assessment
Change from baseline in CDAI score | Baseline up to 24 months
  Measured by investigator assessment
Change from baseline in SDAI score | Baseline up to 24 months
  Measured by investigator assessment
Change from baseline in RAPID3 score | Baseline up to 24 months
  Measured by investigator assessment
Change from baseline in Tender Joint Count of 28 joints (TJC28) score | Baseline up to 24 months
  Measured by patient assessment
Change from baseline in Swollen Joint Count of 28 joints (SJC28) score | Baseline up to 24 months
  Measured by patient assessment
Change from baseline in HAQ-DI score | Baseline up to 24 months
  Measured by patient assessment
Change from baseline in Work Productivity and Activity Impairment (WPAI) score | Baseline up to 24 months
  Measured by patient assessment
Change from baseline in Patient Pain | Baseline up to 24 months
  Measured by patient assessment
Change from baseline in Patient Fatigue | Baseline up to 24 months
  Measured by patient assessment
Number of patients continuing treatment | At 12 months
  Measured by investigator assessment
Number of patients continuing treatment | At 24 months
  Measured by investigator assessment
Number of changes to Rheumatoid Arthritis (RA) treatment | Up to 24 months
  Measured by investigator assessment
Distribution of reasons for changes to Rheumatoid Arthritis (RA) treatment | Up to 12 months
  Measured by questionnaire
Incidence of treatment-emergent Adverse Events | Up to 24 months
  Measured by investigator assessment
Time to achieve sustained CDAI LDA | Up to 12 Months
  Time to achieve sustained Clinical Disease Activity Index (CDAI) Low Disease Activity (LDA)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Westmount, Quebec, Canada

REFERENCES:
- [Derived] Bessette L, Haraoui B, Rampakakis E, Dembowy J, Trepanier MO, Pope J. Effectiveness of a treat-to-target strategy in patients with moderate to severely active rheumatoid arthritis treated with abatacept. Arthritis Res Ther. 2023 Sep 28;25(1):183. doi: 10.1186/s13075-023-03151-2. PMID 37759330
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm